CLINICAL TRIAL: NCT06417008
Title: A Phase Ib/III Clinical Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Immunogenicity of HS-20117 Combined With Aumolertinib in Participants With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of HS-20117 Combined With Aumolertinib in Participants With Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20117-301
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; HS-20117; Epidermal Growth Factor Receptor; c-Mesenchymal-Epithelial Transition; Bispecific Antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ib: HS-20117 and Aumolertinib (Experimental): Participants will receive IV infusion of HS-20117 once during cycle 1 and once every 2 weeks during subsequent cycles (The duration of each treatment cycle is 28 days) at exploratory doses. Aumolertinib will be administered 110 mg orally once daily.
  Interventions: Drug: HS-20117; Drug: Aumolertinib
- Phase III: HS-20117 and Aumolertinib (Experimental): Participants will receive IV infusion of HS-20117 once during cycle 1 and once every 2 weeks during subsequent cycles (The duration of each treatment cycle is 28 days) at exploratory doses. Aumolertinib will be administered 110 mg orally once daily.
  Interventions: Drug: HS-20117; Drug: Aumolertinib
- Phase III: Aumolertinib (Active Comparator): Participants will receive Aumolertinib 110 mg orally once daily.
  Interventions: Drug: Aumolertinib

INTERVENTIONS:
Drug: HS-20117 — Participants will receive HS-20117 once during cycle 1 and once every 2 weeks during subsequent cycles (The duration of each treatment cycle is 28 days)
  Other Names: PM1080
  Arms: Phase III: HS-20117 and Aumolertinib; Phase Ib: HS-20117 and Aumolertinib
Drug: Aumolertinib — 110 mg orally once daily.
  Other Names: Almonertinib Mesilate Tablets; HS-10296; Almonertinib

SUMMARY:
HS-20117 is a fully-human EGFR-MET immunoglobulin G1(IgG1)-like bispecific antibody. The purpose of this study is to assess the safety, efficacy, pharmacokinetics and immunogenicity of HS-20117 combined with Aumolertinib in participants with epidermal growth factor receptor (EGFR) mutation (Exon 19 deletions [Exon 19del] or Exon 21 L858R substitution) positive, locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a multicenter Phase Ib/III clinical study evaluating the safety, efficacy, pharmacokinetics (PK), and immunogenicity of HS-20117 in combination with aumolertinib in subjects with locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC). The study is divided into two phases, Phase Ib, a dose expansion study and Phase III, a confirmatory study. In the dose expansion phase (Phase Ib), HS-20117 will first be studied in combination with the standard dose of aumolertinib, to assess the efficacy, safety, tolerability, PK profile, and immunogenicity of HS-20117 in combination with aumolertinib in the target population, as well as to determine the recommended Phase III dose (RP3D). Following confirmation of the safety and efficacy of HS-20117 in combination with aumolertinib and RP3D in Phase Ib, a randomized, active-controlled, open-label, multicenter Phase III study will be initiated to assess the efficacy and safety of HS-20117 in combination with aumolertinib versus aumolertinib in the target population in the confirmatory study phase.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 - 75 years (inclusive).
* Participants with newly diagnosed histologically or cytologically confirmed, locally advanced or metastatic EGFR-sensitive mutated NSCLC (stage IIIB/IIIC/IV) that is treatment naive and not amenable to curative therapy including surgical resection or chemoradiation.
* Agree to provide fresh or archival tumor tissue.
* At least one target lesion per the RECIST v1.1.
* ECOG performance status of 0-1.
* Minimum life expectancy > 12 weeks.
* Males or Females should be using adequate contraceptive measures throughout the study.
* Females must not be pregnant at screening or have evidence of non-childbearing potential.
* Have signed Informed Consent Form.

Exclusion Criteria:

* Received or are receiving the following treatments:

  1. Previous or current treatment with MET targeted therapy or EGFR targeted antibodies or antibody-drug conjugates (ADC).
  2. Traditional Chinese medicine indicated for tumors, major surgery or other local therapy within washout period to the first dose of study drug.
  3. Presence of pleural effusion/ascites requiring clinical intervention; presence of pericardial effusion.
  4. Other investigational non-anti-tumor drugs, strong CYP3A4 inhibitors, strong inducers, drugs that are sensitive substrates of BCRP or P-gp, or drugs that prolong the QT interval within the washout period.
* Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
* History of other primary malignancies.
* Untreated, or active central nervous system metastases.
* Inadequate bone marrow reserve or organ functions.
* Severe, uncontrolled or active cardiovascular disorders.
* Severe or uncontrolled systemic diseases.
* Severe bleeding symptoms or bleeding tendencies.
* Severe arteriovenous thrombosis occurred.
* Serious or active infection.
* Active infectious diseases.
* Interstitial lung disease (ILD).
* Serious neurological or mental disorders.
* History of hypersensitivity to any component of HS-20117 and Aumolertinib or their similar drugs.
* Female subjects who are pregnant, lactating, or planning to become pregnant or breastfeed during the study period or within 6 months after the last dose of the study drug.
* Subjects with a history of severe allergic reactions or those who have experienced severe infusion reactions
* Participants with any condition that compromises the safety of the participant or interferes with the assessment of the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
[Phase Ib] Objective response rate (ORR) According to response evaluation criteria in solid tumors (RECIST) v1.1 by Investigators (INVs) | From the date of first dose until the date of disease progression or withdrawal from study, up to approximately 40 months
  ORR is defined as the percentage of participants with DOR of confirmed CR or confirmed PR per RECIST v1.1
[Phase III] Progression-Free Survival (PFS) According to RECIST v1.1 by Independent Review Committee(IRC) | Up to approximately 40 months
  PFS is defined as the time from randomization until the date of objective disease progression or death, whichever occurred first, based on IRC using RECIST v1.1

SECONDARY OUTCOMES:
[Phase Ib and III] Overall Survival (OS) | Approximately 60 months
  Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.
[Phase Ib and III] Disease control rate (DCR) According to RECIST v1.1 by INVs | From the date of first dose until the date of disease progression or withdrawal from study, approximately 40 months.
  DCR is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks) based on Investigator's assessment per RECIST v1.1.
[Phase Ib and III] Duration of response (DoR) According to RECIST v1.1 by INVs | From the date of CR, PR until the date of disease progression or death, approximately 40 months.
  DoR only applies to participants whose best overall response is CR or PR based on Investigator's assessment per RECIST v1.1. The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying disease.
[Phase Ib and III] Progression-Free Survival (PFS) According to RECIST v1.1 by INVs | Up to approximately 40 months
  PFS is defined as the time from randomization until the date of objective disease progression or death, whichever occurred first, based on IRC using RECIST v1.1
[Phase III] ORR According to RECIST v1.1 by INVs | From the date of first dose until the date of disease progression or withdrawal from study, up to approximately 40 months
  ORR is defined as the percentage of participants with BOR of CR or PR per RECIST v1.1
[Phase III] ORR According to RECIST v1.1 by IRC | From the date of first dose until the date of disease progression or withdrawal from study, up to approximately 40 months
  ORR is defined as the percentage of participants with BOR of CR or PR per RECIST v1.1
[Phase III] DCR According to RECIST v1.1 by IRC | From the date of first dose until the date of disease progression or withdrawal from study, approximately 40 months.
  DCR is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks)
[Phase III] DoR According to RECIST v1.1 by IRC | From the date of CR, PR until the date of disease progression or death, approximately 40 months.
  DoR only applies to participants whose best overall response is CR or PR. The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying disease.
[Phase Ib and III] Incidence and severity of treatment-emergent adverse events | From the date of first dose until 90 days after the final dose. A cycle is 28 days.
  Adverse event (assessed according to NCI CTCAE v5.0) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
[Phase Ib and III] Immunogenicity of HS-20117 | Cycle 1 Day 1: predose through EOT or follow up period (90 days after the last dose).
  Immunogenicity will be measured by the number of participants that are ADA positive.
[Phase Ib] PK parameters: Maximum serum concentration (Cmax) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The Cmax is the maximum observed serum concentration of HS-20117
[Phase Ib] PK parameters: Trough serum concentration (Ctrough) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  Ctrough is the observed serum concentration immediately prior to the next administration
[Phase Ib] PK parameters: Area under the curve from time Zero to end of dosing interval (AUCtau) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days
  The AUCtau is defined as the area under the serum concentration-time curve during a dose interval time period(tau)
[Phase Ib] PK parameters: Time to reach maximum observed serum concentration (Tmax) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The Tmax is defined as time to reach maximum observed serum concentration of HS-20117
[Phase Ib] PK parameters: Terminal elimination half-life (t1/2) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The t1/2 is defined as the time it takes for the concentration levels to fall to 50% of their value.

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Yun Fan, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang